CLINICAL TRIAL: NCT06341933
Title: Risk Factors for Acute Kidney Injury in Patients Undergoing Video-Assisted Thoracoscopic Surgery for Pulmonary Resection: A Prospective Observational Study
Brief Title: Risk Factors for AKI in Patients Undergoing VATS for Pulmonary Resection
Status: Recruiting | Type: Observational
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Alagoz, Department of anesthesiology and reanimation, Principal Investigator, Specialist Doctor, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Other Study IDs: 2024-BÇEK/41
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Acute Kidney Injury; Surgery; Lung Cancer
Keywords: Acute Kidney Injury; Lung Cancer; Video Assisted Thoracoscopic Surgery
MeSH Terms: conditions — Acute Kidney Injury; Lung Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Acute Kidney Injury (NO): In the postoperative period, patients with normal renal function.
  Interventions: Other: Duration of Surgery; Other: Volume of Fluid in Surgery; Other: Blood Loss
- Acute Kidney Injury (YES): There has been a decrease of more than 25% in the estimated glomerular filtration rate (t-GFH), and/or a 1.5-fold increase in serum creatinine, and/or a 6-hour urine volume of less than 0.5 ml/kg/h.
  Interventions: Other: Duration of Surgery; Other: Volume of Fluid in Surgery; Other: Blood Loss

INTERVENTIONS:
Other: Duration of Surgery — Total surgery time in minutes
Other: Volume of Fluid in Surgery — Fluid volume given during surgery in ml
Other: Blood Loss — Blood loss during surgery in ml

SUMMARY:
This study aims to investigate the potential factors contributing to the development of Acute Kidney Injury (AKI) in patients undergoing pulmonary resection with Video Assisted Thoracoscopic Surgery (VATS) for lung malignancy. The study will focus on demographic data, laboratory parameters, perioperative fluid management, and haemodynamics.

The research will be conducted at SBÜ Ankara Atatürk Sanatorium Training and Research Hospital. The study will involve patients who have given informed consent and will undergo VATS with standard anaesthesia monitoring. Anaesthesia management will follow our routine protocol in our clinic.

Patients will be divided into two groups based on whether they have a more than 25% decrease in estimated glomerular filtration rate (t-GFH) and/or a 1.5-fold increase in serum creatinine and/or a 6-hour urine volume of less than 0.5 ml/kg/h. The patients will be divided into two groups based on this definition, and the risk factors between these groups will be analysed.

The preoperative routine blood values, demographic data (age, gender, height, weight, and BMI), ASA physical status, smoking and alcohol habits, comorbidities, and regular medication use will be recorded. Intraoperative urine output and haemodynamic parameters will also be monitored. Routine blood gas analysis, blood urea nitrogen (BUN), glomerular filtration rate (GFR), albumin, haemoglobin, sodium, potassium, chlorine, and magnesium will be measured and recorded, along with urine output and t-GFH. Patients will be evaluated in the hospital on the day the surgeon calls for a postoperative check-up and on the 30th postoperative day to see if there are any complications.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age, under 65 years of age,
* American Society of Anesthesiologists (ASA) physical status 1-3,
* Data of patients who will undergo wedge resection, segmentectomy or lobectomy with elective VATS due to lung malignancy will be examined prospectively.

Exclusion Criteria:

* Patients with a body mass index (BMI) less than 18.5kg/m2 or greater than 35 kg/m2,
* Those with impaired renal function (the upper limit of the creatinine reference range is more than 50%; 1.3 mg/dL for men and 1.1 mg/dL for women),
* A radiological examination was performed using radiocontrast material in the preoperative period,
* Clinically and radiologically diagnosed with congestive heart failure and treatment has been started,
* Having a history of pulmonary edema,
* Those who have used steroids and non-steroidal anti-inflammatory drugs for a long time (exceeding 30 days),
* Intubated to intensive care unit,
* In need of massive peroperative blood transfusion,
* Patients with deficiencies in the parameters examined will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the given parameters of a 1/3 patient ratio, two-sided (two-tailed) type I error of 0.05, power of 95%, effect size of 0.86, and group distribution ratio of 3, it was determined that the group with acute kidney injury should include 24 patients and the group without acute kidney injury should include 72 patients. Our study was designed to include an average of 100 patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Glomerular Filtration Rate | 1 day
  Glomerular filtration rate (GFR) is the volume of fluid filtered from the renal (kidney) glomerular capillaries into the Bowman's capsule per unit time.
Serum Creatinine | 1 day
  The creatinine blood test measures the level of creatinine in the blood. This test is done to see how well your kidneys are working. Creatinine in the urine can be measured with a urine test. A measurement of the serum creatinine level is often used to evaluate kidney function.
Amount of Urine | 1 day
  The amount of urine produced per hour according to the patient's weight

CONTACTS AND LOCATIONS:
Overall Officials: Ali ALAGÖZ, professor, Principal Investigator — Ankara Ataturk Sanatorium Training and Research Hospital
Locations (1):
- Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No